CLINICAL TRIAL: NCT07250971
Title: Efficacy of Virtual Reality-Based Psychotherapeutic and Psychoeducational Interventions on Anxiety and Depression Symptoms
Brief Title: Virtual Reality-Based Psychotherapeutic and Psychoeducational Intervention for Anxiety and Depression in Children, Adolescents, and Adults
Acronym: VR-PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, Çağlar Charles Daniel Jaicks, Assist. Prof. Dr., Istanbul Aydın University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAU-VR-160-2025; 160/2025 (Other: Non-Interventional Clinical Research Ethics Committee of Istanbul Aydın University)
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Anxiety Disorders; Depressive Disorders
Keywords: Virtual Reality; Psychotherapy; Psychoeducation; Non-Pharmacological Treatment; Mental Health; Adolescents; Depression; Anxiety; Digital Therapeutics; Immersive Therapy
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Psychological Well-Being; Depression

STUDY DESIGN:
Intervention Model Description: All participants received the same virtual reality (VR)-based psychotherapeutic and psychoeducational intervention consisting of five weekly sessions. Each session included relaxation, exposure, coping skills, and psychoeducation modules delivered through Meta Quest 2 headsets under professional supervision. There were no control or comparison groups. A pre-test-post-test design was used to measure changes in anxiety and depression symptoms before and after the VR intervention.
Masking Description: This study was conducted as an open-label design. Neither participants nor investigators were blinded to the intervention. All participants received the same virtual reality (VR)-based psychotherapeutic and psychoeducational sessions, and both the participants and supervising clinicians were fully aware of the intervention content and duration. No masking procedures were implemented, as the behavioral nature of the study required active participant engagement with the VR program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality-Based Psychotherapeutic and Psychoeducational Intervention (Experimental): All participants received a virtual reality (VR)-based psychotherapeutic and psychoeducational program consisting of five weekly individual sessions lasting 20-40 minutes each. The intervention included modules on relaxation and breathing exercises, exposure, coping strategies, study skills, and sleep hygiene. Sessions were delivered using Meta Quest 2 headsets under professional supervision.
  Interventions: Behavioral: Virtual Reality-Based Psychotherapeutic Program

INTERVENTIONS:
Behavioral: Virtual Reality-Based Psychotherapeutic Program — A behavioral intervention delivered through virtual reality (VR) technology designed to reduce symptoms of anxiety and depression. The program included immersive psychoeducational and psychotherapeutic content focusing on relaxation, exposure, coping skills, and healthy routines. Each participant completed five supervised weekly sessions using Meta Quest 2 headsets.

SUMMARY:
This study is designed as a non-pharmacological, interventional clinical research project to evaluate the feasibility, safety, and implementation of virtual reality (VR)-based psychoeducational and psychotherapeutic interventions for individuals with anxiety and/or depression. Participants include children, adolescents, and adults who meet DSM-5 diagnostic criteria or present with subthreshold symptoms associated with functional impairment and who decline pharmacological treatment.

A total of 40 participants are planned to receive five weekly individual VR sessions conducted under the supervision of a psychiatrist or clinical psychologist. The VR intervention will be administered using Meta Quest 2 headsets and will include modules focused on relaxation and breathing exercises, exposure-based tasks, coping strategies for anxiety and procrastination, study skills (e.g., Pomodoro technique), sleep hygiene, and psychoeducation about healthy behaviors. Each session will last approximately 20-40 minutes and will be conducted in a controlled clinical environment to ensure participant safety.

Anxiety and depression levels will be assessed before and after the intervention using validated clinical scales, including the Hamilton Depression Rating Scale and the Beck Depression Inventory. Side effects such as dizziness, nausea, and disorientation will be monitored throughout the study. The primary objective is to evaluate feasibility, implementation, and acceptability of VR-based interventions in a clinical mental health setting. Secondary objectives include exploring pre-post changes in anxiety and depression scores and documenting safety and tolerability of the VR intervention.

DETAILED DESCRIPTION:
This study is designed as a non-pharmacological, interventional clinical research project to evaluate the feasibility, safety, and implementation of virtual reality (VR)-based psychoeducational and psychotherapeutic interventions for individuals with anxiety and/or depression. Participants include children, adolescents, and adults who meet DSM-5 diagnostic criteria or present with subthreshold symptoms associated with functional impairment and who decline pharmacological treatment.

A total of 40 participants are planned to receive five weekly individual VR sessions conducted under the supervision of a psychiatrist or clinical psychologist. The VR intervention will be administered using Meta Quest 2 headsets and will include modules focused on relaxation and breathing exercises, exposure-based tasks, coping strategies for anxiety and procrastination, study skills (e.g., Pomodoro technique), sleep hygiene, and psychoeducation about healthy behaviors. Each session will last approximately 20-40 minutes and will be conducted in a controlled clinical environment to ensure participant safety.

Anxiety and depression levels will be assessed before and after the intervention using validated clinical scales, including the Hamilton Depression Rating Scale and the Beck Depression Inventory. Side effects such as dizziness, nausea, and disorientation will be monitored throughout the study. The primary objective is to evaluate feasibility, implementation, and acceptability of VR-based interventions in a clinical mental health setting. Secondary objectives include exploring pre-post changes in anxiety and depression scores and documenting safety and tolerability of the VR intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of anxiety and/or depression according to DSM-5 criteria, or presence of subthreshold symptoms associated with functional impairment.
* Age between 12 and 25 years.
* No psychopharmacological treatment within the past 12 months.
* Voluntary participation and written informed consent for the virtual reality sessions.
* Sufficient cognitive capacity to understand and engage with VR-based interventions.
* Referred by a qualified mental health professional for non-pharmacological therapy.

Exclusion Criteria:

* History of epilepsy, hypertension, or neurological/cardiovascular conditions that contraindicate the use of virtual reality.
* Presence of psychotic disorder or severe cognitive impairment.
* Stent placement in cerebral or cardiac vessels.
* Current or past-year use of psychiatric medication.
* Refusal or inability to tolerate virtual reality exposure.
* Any medical or psychiatric condition that prevents safe participation in VR sessions.

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2025-07-09 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change in Depression Severity Measured by Hamilton Depression Rating Scale (HAM-D) | Baseline and Week 5 (end of intervention)
  Depression severity will be measured using the Hamilton Depression Rating Scale (HAM-D) before and after completion of the five-session VR intervention. The total score ranges from 0 to 52, with higher scores indicating greater depressive symptom severity. A decrease in total score represents clinical improvement.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Aydın University, Department of Child and Adolescent Psychiatry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy and ethical considerations involving sensitive mental health information.